CLINICAL TRIAL: NCT02522481
Title: A Prospective Multicenter Phase III Clinical Evaluation of the Safety and Efficacy of Lumason™/SonoVue® in Subjects Undergoing Pharmacologic Stress Echocardiography With Dobutamine for the Diagnosis of Coronary Artery Disease
Brief Title: Evaluation of Safety and Efficacy of Lumason/SonoVue in Subjects Undergoing Pharmacologic Stress BR1-141
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR1-141
Record Dates: First submitted 2015-07-17; First posted 2015-08-13 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: Lumason; Dobutamine stress echo; stress echo; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lumason (Experimental): Lumason (sulfur hexafluoride lipid-type A microspheres) 2 mL IV injection
  Interventions: Drug: Lumason

INTERVENTIONS:
Drug: Lumason — Lumason (sulfur hexafluoride-type A microspheres) an ultrasound contrast agent was administered as 2 single 2-mL IV injections during rest and stress echocardiography
  Other Names: SonoVue

SUMMARY:
The purpose of this study was to assess the safety and efficacy of Lumason-enhanced dobutamine stress echo (CE-DSE) in subjects having a suboptimal left ventricular endocardial border delineation (LV EBD) at rest and who were scheduled for coronary angiography.

DETAILED DESCRIPTION:
The study was designed to assess the safety and efficacy of Lumason at improving the visualization of the LV EBD during pharmacologic stress echocardiography examinations and for detection or exclusion of the coronary artery disease (CAD). The study population consisted of adult subjects referred for pharmacological stress echocardiography and with suboptimal image quality during unenhanced ultrasound imaging at rest who had known or suspected CAD. Subjects enrolled in the study represented subjects who could benefit most from contrast-enhanced ultrasound (CEUS) stress echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Provided written Informed Consent and was willing to comply with protocol requirements;
* Was at least 18 years of age;
* Had suspected or known CAD and was scheduled to undergo coronary angiography within 6 months after the LUMASON DSE.
* Had undergone a previous echocardiography prior to enrollment; resulting in suboptimal unenhanced images at rest, defined as ≥ 2 suboptimal adjacent segments in any apical view.

Exclusion Criteria:

* Was a pregnant or lactating female. Excluded the possibility of pregnancy by testing on site at the institution (serum or urine βHCG) within 24 hours prior to the start of LUMASON administration(s), by surgical history (e.g., tubal ligation or hysterectomy), post menopausal with a minimum 1 year without menses;
* Had any known hypersensitivity to 1 or more ingredients of LUMASON (sulfur hexafluoride or to any components of LUMASON);
* Had any known hypersensitivity to dobutamine;
* Had an ongoing or recent (within the last 30 days) acute myocardial infarction;
* Had known right-to-left, bidirectional or transient cardiac shunt (ruled out with agitated saline study performed before administration of LUMASON);
* Had electrolyte (especially potassium and magnesium) abnormalities;
* Had unstable pulmonary and/or systemic hemodynamic conditions e.g.:
* decompensated or inadequately controlled congestive heart failure (NYHA Class IV);
* hypovolemia;
* uncontrolled hypertension, i.e. resting systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg;
* unstable angina;
* acute coronary syndrome;
* aortic dissection;
* acute pericarditis,
* myocarditis, or endocarditis;
* stenosis of the main left coronary artery;
* hemodynamically significant outflow obstruction of the left ventricle, including hypertrophic obstructive cardiomyopathy;
* hemodynamically significant cardiac valvular defect;
* acute pulmonary embolism;
* Had uncontrolled cardiac arrhythmias;
* Had significant disturbance in conduction;
* Had hypertrophic subaortic stenosis;
* Had an acute illness (e.g., infections, hyperthyroidism, or severe anemia);
* Was previously entered into this study or received an investigational compound within 30 days before admission into this study;
* Had been treated with any other contrast agent either intravascularly or orally within 48 hours of the first LUMASON administration;
* Had any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or postdose follow-up examinations;

In addition, due to the use of Atropine in subjects who had not reached targeted heart rate with peak dobutamine infusion, subjects with the following were excluded:

* Glaucoma;
* Pyloric stenosis;
* Prostatic hypertrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2018-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melda Dolan, MD, Study Director — Bracco Diagnostics, Inc
Locations (17):
- United States (10):
  - Sarver Heart Center, University of Arizona, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - Interventional Cardiology Medical Group, Inc., West Hills, California
  - Cardiology Physicians, PA, Newark, Delaware
  - Community Heart and Vascular Community Hospital East, Indianapolis, Indiana
  - St. Luke's Mid-America Heart Institute, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - The Institute for Clinical Research Holy Name Medical Center, Teaneck, New Jersey
  - Mount Sinai Medical Center, New York, New York
- Mazankowski Alberta Heart Institute, University of Alberta Hospital, Edmonton, Alberta, Canada
- Germany (4):
  - Medizinische Klinik m.S. Kardiologie und Angiologie, Charité Universitätsmedizin Berlin, Berlin
  - Klinikum Lünen, St. Marien-Hospital GmbH, Lünen
  - Universitätsmedizin Mainz, Mainz
  - Kardiologie Klinik Dr. Müller GmbH, Peter Osypka Heart Center, Munich
- Italy (2):
  - Azienda Ospedaliera Universitaria Parma, Parma
  - Azienda Policlinico Umberto I Università degli Studi di Roma La Sapienza, Rome

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumason
Started | 175
Completed | 172
Not Completed | 3
Not completed — discontinued | 1
Not completed — Not dosed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lumason
Number analyzed (Participants) | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 160
  More than one race | 4
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.33 (7.252)
Height [Mean (Standard Deviation); unit: cm] | 169.3 (10.49)
Weight [Mean (Standard Deviation); unit: kg] | 86.99 (21.781)

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity for Detection or Exclusion of Coronary Artery Disease (CAD)
Description: The diagnostic performance of the echocardiographic images was compared to the truth standard to determine sensitivity and specificity. A diagnosis of coronary artery disease (CAD) was determined for both the echo images and truth standard (positive diagnosis for CAD is defined as >/= 50% stenosis of any vessel on coronary angiography or if no coronary angiography is performed the occurence of a cardiac event based on clinical information for up to 6 months post dose; otherwise the diagnosis is negative).
  Results for sensitivity and specificity are reflected based on difference between contrast enhanced stress echo and unenhanced stress echo. Results for analysis of data based on majority assessment from the three off-site blinded readers are presented.
  Sensitivity and specificity are the percentages of correctly diagnosed subjects by stress echo over the total positive and negative subjects according to the truth standard respectively.
Time Frame: Participants were followed until they had coronary angiography or up to 6 months post dose to collect clinical information on cardiac events if no coronary angiography were performed
Population: Analysis population for coronary artery disease (CAD) included all subjects who received Lumason, had overall diagnostic conclusion of CAD available at peak stress for both UE-DSE and CE-DSE and had a definite truth standard diagnosis (Positive, Negative) for CAD (coronary angiography or 6 months collection of cardiac events follow-up data).
Measure: Number; unit: percentage of participants
Groups:
- CE-DSE - UE-DSE: Difference between contrast-enhanced dobutamine stress echo (CE-DSE) and unenhanced dobutamine stress echo (UE-DSE) (CE-DSE - UE-DSE)
Arm/Group | CE-DSE - UE-DSE
Number analyzed (Participants) | 170
percentage of participants
  Sensitivity | 8.0
  Specificity | 33.7
Statistical Analysis 1: Comparison: CE-DSE - UE-DSE; Sensitivity: superiority test comparing CE-DSE and UE-DSE based on the difference; Test type: Superiority; p = 0.0896, McNemar
Statistical Analysis 2: Comparison: CE-DSE - UE-DSE; Specificity: superiority test comparing CE-DSE and UE-DSE based on the difference; Test type: Superiority; p < 0.0001, McNemar

2. Primary Outcome: Reader-Specific Percentages of Participants Identified as Having a Critical Shift From Suboptimal to Optimal Echocardiographic Images
Description: The percentage of subjects with suboptimal images (defined as >= 2 adjacent segments with inadequate left ventricular endocardial border delineation (LV EBD) in any of the 3 apical views) at unenhanced stress echo converted to adequate (reduction of suboptimal segments in any of the 3 apical views) at contrast-enhanced stress echo
Time Frame: Participants were followed until they had coronary angiography or up to 6 months post dose to collect clinical information on cardiac events if no coronary angiography was performed
Population: The analysis population for EBD included all subjects who received Lumason and had EBD data available at peak stress for both UE-DSE and CE-DSE.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Reader 1: Reader 1 CE-DSE
- Reader 2: Reader 2 CE-DSE
- Reader 3: Reader 3 CE-DSE
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 167 | 167 | 167
percentage of participants | 84.4 [74.4 to 91.7] | 93.7 [87.9 to 97.2] | 78.8 [67.0 to 87.9]

3. Secondary Outcome: Change in Total LV EBD
Description: Measured as the change in the total LV EBD score based on the 17 segments, from peak stress unenhanced vs. peak stress contrast-enhanced. Total LV EBD score ranges from 0 to 34 and higher score is better outcome.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- UE-DSE: Unenhanced DSE
- CE-DSE: Contrast-enhanced DSE
- Difference: (CE-DSE - UE-DSE)
Arm/Group | UE-DSE | CE-DSE | Difference
Number analyzed (Participants) | 167 | 167 | 167
score on a scale
  Reader 1 | 17.5 (10.83) | 28.1 (8.32) | 10.6 (11.98)
  Reader 2 | 13.4 (8.57) | 30.5 (4.81) | 17.1 (7.87)
  Reader 3 | 17.8 (7.04) | 23.6 (7.47) | 5.8 (9.17)

4. Secondary Outcome: Number of Participants With Adverse Events
Description: To obtain safety data in subjects administered Lumason during echocardiography
Time Frame: up to 72 hours post dose
Population: Safety analysis population includes all subjects who received Lumason
Measure: Number; unit: participants
Groups:
- Lumason: All patients were administered, Lumason (sulphur hexafluoride lipid-type A microspheres) an ultrasound contrast agent as a single 0.03 mL/kg bolus injection during echocardiography
Arm/Group | Lumason
Number analyzed (Participants) | 173
participants
  Number of subjects with adverse events (AE) | 21
  Number of subjects with AEs by intensity - Mild | 15
  Number of subjects with AEs by intensity -Moderate | 5
  Number of subjects with AEs by intensity - Severe | 1
  Number of subjects with serious AEs | 3

ADVERSE EVENTS:
Time Frame: All adverse events (AE) that occurred from the time the subject signed the Informed Consent Form (ICF) until 72 hours after the last administration of Lumason or until the subject underwent cardiac intervention, whichever came first, were listed [recorded], [with predose AEs flagged in the subject data listings.]
Arm/Group | Lumason
All-Cause Mortality (participants affected / at risk) | 0/173
Serious Adverse Events (participants affected / at risk) | 3/173
Other Adverse Events (participants affected / at risk) | 21/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumason (N=173)
phlebitis (Vascular disorders) | 1 (1)
acute myocardial infarction (Cardiac disorders) | 1 (1)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumason (N=173)
Bifascicular block (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Electrocardiogram change (Investigations) | 1 (1)
Haematocrit increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT02522481/Prot_SAP_000.pdf